CLINICAL TRIAL: NCT05906693
Title: A Cross-sectional Study - The Quality of Life in Individuals With Parkinson's Disease: Is it Related to Functionality and Tremor Severity?
Brief Title: The Quality of Life in Individuals With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Buse KILINÇ, PT.MSc., Pamukkale University
Other Study IDs: 60116787-020/45991; 2019SABE021 (Other Grant/Funding Number: PAU Scientific Research Projects Coordination)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Tremor; Functionality
Keywords: Quality of Life; Upper Limb Functionality; Tremor; Electromyography; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Quality of Life; Hand Strength; Pinch Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life — Parkinson's Disease Quality of Life Questionnaire (PDQ-39)
Other: Upper limb functionality — Nine-Hole Peg Test
Other: Grip and pinch strength — Dynamometer
Other: Tremor amplitude — Electromyography
Other: Depression and anxiety levels — Hospital Anxiety and Depression Scale
Other: Clinical manifestations — The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale

SUMMARY:
This study aimed to examine the relationship of quality of life with tremor severity and upper limb functionality in individuals with Parkinson's Disease. The differences between Parkinson's Disease Quality of Life Questionnaire, Nine-Hole Peg Test, grip and pinch strength values in the individuals with and without tremor in the study were investigated.

DETAILED DESCRIPTION:
Evaluating the relationship between Quality of Life and tremor is needed to determine the best physiotherapy and rehabilitation approaches for individuals with Parkinson's Disease. This study aimed to examine the relationship of quality of life with tremor severity and upper limb functionality in individuals with Parkinson's Disease. Fifty-two individuals with Parkinson's Disease participated in the study. Quality of Life, tremor amplitude, upper limb functionality, grip and pinch strength were evaluated. The relationship of quality of life with tremor severity and upper limb functionality was examined in individuals with Parkinson's Disease. The results of individuals with and without tremor were compared.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of idiopathic Parkinson Disease
* Age between 40 and 80 years
* Being literate
* Having a grade between 1-4 from the Modified Hoehn and Yahr Scale
* Having a score lower than 11 in Hospital Anxiety and Depression Scale

Exclusion Criteria:

* Who were with any other neurologic or orthopedic or rheumatologic disease affecting the upper extremity
* Using antidepressants
* Having vision loss
* Deep brain stimulation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson Disease were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale | 1 year
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale. Used for the evaluation of clinical manifestations of Parkinson's disease. The scale consists of 4 subscales: the first part is Non-Motor Aspects of Experiences of Daily Living (13), the second part is Motor Aspects of Experiences of Daily Living (13), the third part is Motor Examination (33), and the fourth part is Motor Complications (6). The total number of items in the scale is 65. The minimum score is 0. The maximum MDS-UPDRS score is higher, given the additional items and scores for each body area, with a maximum score of 272. Higher scores indicate greater impact of Parkinson Disease symptoms.
Hospital Anxiety and Depression Scale | 1 year
  The Hospital Anxiety and Depression Scale aims to measure symptoms of anxiety and depression and consists of 14 items, seven items for the anxiety subscale (Hospital Anxiety and Depression Scale Anxiety) and seven for the depression subscale (Hospital Anxiety and Depression Scale Depression). Each item is scored on a response-scale with four alternatives ranging between 0 and 3. After adjusting for six items that are reversed scored, all responses are summed to obtain the two subscales. Both depression and anxiety subheadings are scored between 0 and 21. Higher scores indicate greater levels of anxiety or depression. Cut-off scores are 8-10 for doubtful cases and ≥11 for definite cases.
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 1 year
  Used to assess the quality of life of Parkinson's patients
Electromyography | 1 year
  Used to assess the tremor amplitude of Parkinson's patients
Nine-Hole Peg Test | 1 year
  Used to assess the upper limb functionality of Parkinson's patients
Dynamometer | 1 year
  Used to assess the grip and pinch strength of Parkinson's patients

CONTACTS AND LOCATIONS:
Overall Officials: Buse KILINÇ, PT.MSc., Principal Investigator — Pamukkale University; Nilüfer ÇETİŞLİ-KORKMAZ, PT.PhD.Prof., Study Director — Pamukkale University; Levent S. BIR, MD.PhD.Prof., Study Chair — Pamukkale University; Ahmet D. MARANGOZ, MD., Study Chair — Klinikum Stuttgart; Hande ŞENOL, Assist.Prof., Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhlman GD, Flanigan JL, Sperling SA, Barrett MJ. Predictors of health-related quality of life in Parkinson's disease. Parkinsonism Relat Disord. 2019 Aug;65:86-90. doi: 10.1016/j.parkreldis.2019.05.009. Epub 2019 May 7. PMID 31118162
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Louis ED, Machado DG. Tremor-related quality of life: A comparison of essential tremor vs. Parkinson's disease patients. Parkinsonism Relat Disord. 2015 Jul;21(7):729-35. doi: 10.1016/j.parkreldis.2015.04.019. Epub 2015 Apr 24. PMID 25952960

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05906693/SAP_000.pdf